CLINICAL TRIAL: NCT05201937
Title: A Phase 1, Open-Label Study in Healthy Adult Participants to Assess the Pharmacokinetics of JNJ-64281802 Administered as Different Multiple Dose Regimens
Brief Title: A Study of JNJ-64281802 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CR109139; 2021-005574-25 (EudraCT Number); 64281802DNG1008 (Other: Janssen Research and development, LLC)
Record Dates: First submitted 2022-01-12; First posted 2022-01-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A: Panel 1 (JNJ-64281802 High Dose Regimen) (Experimental): Participants will receive Loading Dose (LD) 1 of JNJ-64281802 twice daily on Days 1 and 2 followed by maintenance Dose (MD) 1 of JNJ-64281802 once daily on Days 3, 10, 17 and 24.
  Interventions: Drug: JNJ-64281802
- Arm A: Panel 2 (JNJ-64281802 High Dose Regimen) (Experimental): Participants will receive LD 1 of JNJ-64281802 twice daily on Days 1 and 2 followed by MD 2 of JNJ-64281802 once daily on Days 3, 6, 10, 13, 17, 20, 24, and 27.
  Interventions: Drug: JNJ-64281802
- Arm B: Panel 3 (JNJ-64281802 Low Dose Regimen) (Experimental): Participants will receive LD 2 of JNJ-64281802 twice daily on Days 1 and 2 followed by MD 3 of JNJ-64281802 once daily on Days 3, 10, 17 and 24.
  Interventions: Drug: JNJ-64281802
- Arm B: Panel 4 (JNJ-64281802 Low Dose Regimen) (Experimental): Participants will receive LD 2 of JNJ-64281802 twice daily on Days 1 and 2 followed by MD 4 of JNJ-64281802 once daily on Days 3, 6, 10, 13, 17, 20, 24, and 27.
  Interventions: Drug: JNJ-64281802
- Arm C: Panel 5 (JNJ-64281802 [Optional]) (Experimental): Participants dosing regimen(s) will be determined based on the results of Study Arm A and Study Arm B.
  Interventions: Drug: JNJ-64281802
- Arm C: Panel 6 (JNJ-64281802 [Optional]) (Experimental): Participants dosing regimen(s) will be determined based on the results of Study Arm A and Study Arm B.
  Interventions: Drug: JNJ-64281802

INTERVENTIONS:
Drug: JNJ-64281802 — JNJ-64281802 tablets will be administered orally as per the defined regimens.

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (PK) of JNJ-64281802 in healthy participants when administered in different multiple dose regimens and as different dose strengths.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history (at screening only), and vital signs performed at screening and Day -1. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study
* Body weight not less than 50 kilogram (kg) and body mass index (BMI) within the range 18.0 and 30.0 kilogram per meter square (kg/m^2), extremes included, at screening and Day -1
* All women must have a negative highly sensitive serum (beta human chorionic gonadotropin [beta hCG]) at screening and a negative urine pregnancy test at Day -1
* Contraceptive use should be consistent with local regulations regarding the use of contraceptive methods for participant participating in clinical studies
* Must sign an informed consent form (ICF) indicating that the participant understands the purpose of, and procedures required for, the study and is willing to participate in the study, before starting any screening activities

Exclusion Criteria:

* Any history of clinically significant skin disease such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Known allergies, hypersensitivity, or intolerance to JNJ-64281802 or its excipients
* Has been dosed with JNJ-64281802 in past 3 months
* Current human immunodeficiency virus type 1 (HIV-1) or type 2 (HIV-2) infection (confirmed by antibodies) at screening
* Current Coronavirus disease 2019 (COVID-19) infection (confirmed by severe acute respiratory syndrome coronavirus 2 [SARS-CoV2] polymerase chain reaction [PCR]) at the time of admission to the study site (Day -1)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2022-12-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of JNJ-64281802 | Up to Day 62
  Cmax is defined as maximum observed plasma concentration of JNJ-64281802.
Time to Reach the Maximum Observed Plasma Concentration (Tmax) of JNJ-64281802 | Up to Day 62
  Tmax is defined the actual sampling time to reach the maximum observed plasma concentration of JNJ-64281802.
Observed Plasma Concentration of JNJ-64281802 Just Prior to the Beginning of a Dosing Interval (Ctrough) | Up to Day 62
  Ctrough is defined as observed plasma concentration of JNJ-64281802 just prior to the beginning of a dosing interval.
Apparent Terminal Elimination Half-life (t1/2) of JNJ-64281802 | Up to Day 62
  t1/2 is defined as apparent terminal elimination half-life of JNJ-64281802.
Area Under the Curve From Time Zero to Last Measurable Concentration (AUC[0-last]) of JNJ-64281802 | Up to Day 62
  AUC(0-last) is defined as area under the curve from time 0 to the time of the last measurable concentration of JNJ-64281802.
Area Under the Curve From Time Zero to Infinity (AUC[0-inf]) of JNJ-64281802 | Up to Day 62
  AUC(0-inf) is defined as area under the curve of JNJ-64281802 from time 0 to infinity time.
Area Under the Curve From Time Zero to tau (AUC[0-tau]) of JNJ-64281802 | Up to Day 62
  AUC(0-tau) is defined as area under the curve from time 0 to tau hours post dose of JNJ-64281802.
Total Apparent Oral Clearance (CL/F) of JNJ-64281802 | Up to Day 62
  CL/F is defined as total apparent oral clearance of JNJ-64281802.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) | Up to 62 days
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Number of Participants with Abnormalities in 12-lead Electrocardiograms (ECGs) | Up to 62 days
  Number of participants with abnormalities in 12-lead ECGs will be reported.
Number of Participants with Abnormalities in Physical Examinations | Up to 62 days
  Number of participants with abnormalities in physical examinations (including skin examination, height and body weight) will be reported.
Number of Participants with Abnormalities in Vital Sign Measurements | Up to 62 days
  Number of participants with abnormalities in vital sign measurements (including temperature, temporal artery measurements, pulse/heart rate and blood pressure) will be reported.
Number of Participants with Abnormalities in Clinical Laboratory Tests | Up to 62 days
  Number of participants with abnormalities in clinical laboratory tests (including hematology, serum chemistry and urinalysis) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- PRA Health Sciences Onderzoekscentrum Groningen, locatie Martini, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency